CLINICAL TRIAL: NCT04076735
Title: DIFFIR: Geriatric Distal Femur Fixation Versus Replacement - A Randomized Controlled Trial of Acute Open Reduction Internal Fixation (ORIF) Versus Distal Femoral Replacement (DFR)
Brief Title: DIFFIR - Geriatric Distal Femur Fixation Versus Replacement
Acronym: DIFFIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); NYU Langone Health (Other); Brigham and Women's Hospital (Other); Queen Elizabeth II Health Sciences Centre (Other); Hamilton Health Sciences Corporation (Other); Yale New Haven Health System Center for Healthcare Solutions (Other); Oregon Health and Science University (Other); OrthoCincy Orthopaedics & Sports Medicine (Unknown); University of California (Other); Hospital for Special Surgery, New York (Other); Stanford University (Other); Cedars-Sinai Medical Center (Other); Thunder Bay Regional Health Sciences Centre (Other); University of California, San Francisco (Other); University of Arkansas (Other); University of Calgary (Other); Ascension Health (Industry); University of Otago (Other); Gold Coast University Hospital, Australia (Unknown); Humber River Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-145
Record Dates: First submitted 2019-08-21; First posted 2019-09-03 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Distal Femur Fracture
Keywords: Distal Femur Fracture; Geriatric fracture
MeSH Terms: conditions — Femoral Fractures, Distal | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized controlled trial comparing acute distal femoral replacement versus surgical fixation as a treatment for geriatric comminuted bi-condylar distal femur fractures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Distal femoral replacement (DFR) (Experimental): Distal femoral replacement will be performed by excising the distal portion of the femur (up to two thirds) and replacing with a prosthesis incorporating a hinged total knee replacement.
  Surgical approach and implant selection will be at the discretion of the treating surgeon and within the standard of care. Surgeons performing this procedure will be qualified by training and experience in arthroplasty.
  Interventions: Procedure: Distal femoral replacement
- Surgical Fixation (ORIF) (Active Comparator): Surgical fixation of the distal femoral fracture will be performed with the goals of obtaining and maintaining anatomic reduction and stable fixation of the distal portion of the femur. Surgical approach and implant selection for the surgical fixation (ORIF) will be at the discretion of the treating surgeon and within the standard of care. Surgeons performing this procedure will be qualified by training and experience in trauma of the knee.
  Interventions: Procedure: Surgical Fixation (ORIF)

INTERVENTIONS:
Procedure: Distal femoral replacement — The distal portion of the femur (up to two thirds) is excised and replaced by a endoprosthesis incorporating a hinged total knee replacement.
  Arms: Distal femoral replacement (DFR)
Procedure: Surgical Fixation (ORIF) — A trained orthopaedic surgeon uses open or minimally invasive reduction techniques and achieves stable fixation with internal fixation devices (plates/screws or intramedullary nail) to restore structural integrity and alignment of the distal femur
  Other Names: open reduction and internal fixation
  Arms: Surgical Fixation (ORIF)

SUMMARY:
The current standard of care for most intra-articular distal femur fractures (above the knee joint) in geriatric patients is a surgical fixation using plates and screws to hold the fracture pieces in the correct position, until the fracture as healed.

However, surgical fixation of these complex fractures in geriatric patients, is associated with significant complications, such as non-union (when the broken bone does not heal properly), infection and the need for revision surgery. Additionally, surgical fixation requires prolonged immobilization of of the affected limb (typically around 6-12 weeks post-operatively), which can lead to disability and other complications. Geriatric patients, especially those frail and with cognition impairment, are unable to adhere to the immobilization restrictions, which leads to an increased risk of fixation failure (broken bone does not heal).

Another treatment option for those patients is an acute distal femoral replacement (artificial knee), where damaged parts of the knee joint are replaced with artificial prosthesis. This procedure allows patients to walk immediately after the surgery and faster return to previous level of function, therefore avoiding the complications for immobilization.

There is a lack of guideline and evidence to suggest which surgical technique is best to provide superior function outcomes, lower complications and reduced costs. The proposed study seeks to answer this question by performing a large clinical trial comparing knee replacement versus surgical fixation in geriatric patients with distal femur fracture.

DETAILED DESCRIPTION:
The proposed study is a prospective, randomized controlled trial, involving multiple centers across North America, to compare distal femur replacement (knee prosthesis) versus surgical fixation as a treatment for geriatric distal femur fracture.

Patients 65 years of age and older, with closed, displaced ( when the two ends of the bone are not lined up straight), comminuted (bone is in many pieces) distal femur fracture, who meet the inclusion criteria and agree to participate in the study, will be randomly assigned (by chance like flipping a coin) to receive either acute distal femoral replacement or surgical fixation.

The hypothesis is that patients in the acute distal femoral replacement group will have superior function, range of motion (full movement potential of a joint), general health status, reduced pain, and lower complications when compared to patients in the surgical fixation group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 65 years and older
* Isolated fracture of the distal femur (Classification 33)
* Fracture is amendable to both treatments
* Fracture is acute (within 2 weeks from time of injury)
* Patient was ambulatory (with or without walking aids) prior to the injury
* Independent or moderately frail with score of 3 to 6 on the Clinical Frailty Scale
* Patient is able to read and understand English, French, or Spanish
* Patient or substitute decision maker is able to provide written informed consent to participate in the study

Exclusion Criteria:

* Active or previous infection around the fracture (soft tissue or bone)
* Open fracture
* Bilateral femur fractures
* Major vascular injuries requiring intervention, compartment syndrome and major neurologic injuries
* Pathological fracture excluding osteoporosis
* Previous surgical fixation or total knee replacement of the distal femur or proximal tibia
* Previous surgical fixation or hemi/total replacement of the hip
* Current or previous extensor mechanism (patellar tendon, quadriceps tendon, or patella fracture) disruption or repair
* Polytrauma (Injury Severity Score > 15) or any associated major injuries of the lower extremities
* Previous medical diagnosis of dementia
* Medical or surgical contra-indication to surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | Our primary outcome is knee pain and function as measured by repeated measures of the Oxford Knee Score at 3, 6, 9 and 12 -months post-surgery to detect a 5 point improvement on the OKS with 0.5 correlation between assessments.
  A short questionnaire consists of 12 questions ranging from 0 to 48 points, designed to assess function and pain after knee replacement surgery. Higher values represent a better outcome. Scores between 40-48 indicate satisfactory joint function.

SECONDARY OUTCOMES:
Daily morphine equivalent usage while in hospital | The outcome will be assessed daily from the day of the surgery until the patient gets discharge from the hospital (24 hours up to 7 days)
  Assess patient's cumulative intake of any drugs in the opioid class (in Milligram Morphine Equivalent) over 24 hours while in hospital.
Visual Analog Pain Scale (VAS) | Pain scale will be assessed immediately after surgery at 24 hours 48 hours, and then at each follow up visit at 3, 6, 9, 12, and 24 months post-surgery
  Assess pain from a visual scale that ranges from 0 to 10. Straight line with the endpoints defining extreme limits such as 'no pain at all' (zero) and 'pain as bad as it could be' (ten)
Health status and quality of life - EQ-5D questionnaire | Questionnaire will be completed by patients at 3, 6, 9, 12, and 24 months post-surgery
  The European Quality of Life 5 Dimensions (EQ5D) is a patient reported outcome where patients self rate their level of severity of health status and health related quality of life. Consists of 5 dimensions (mobility, selfcare, usual activities, pain/discomfort, anxiety/depression) and each one of them has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) where patients will indicate how they feel regarding their health status and quality of life.
knee range of movement (ROM) | Test will be completed at each follow up visit at 3, 6,12 and 24 months post surgery
  The therapist/assessor uses a goniometer (instrument that measures an angle of a joint) to measure the degree of knee flexion and extension of a patient.
  Knee Flexion - the measurable degree in which the leg (and knee joint) is bent. Knee Extension - The measurable degree in which the knee is extended (making the joint angle larger, or straightening the knee)
Timed Up and Go (TUG) test | Test will be completed at each follow up visit at 3, 6, 12 and 24 months post surgery
  TUG is a simple test used to assess a person's mobility (in seconds) and requires both static and dynamic balance. A line is placed on the floor 3 meters away from a chair where patient will be sitting.
  When instructed to "GO" patient will stand, walk to a line on the floor at his/her regular pace, turn around and walk back to the chair and sit down. The longer it takes for subject to complete the test, higher is the risk of fall and lower is the its functional mobility.
  Reference values are:
  60-69 years old = 8.1 seconds; 70-79 years old = 9.2 seconds; 80-99 years old = 11.3 seconds. Over 14 seconds is associate with high risk of fall
Knee Extension lag | Test will be completed at each follow up visit at 3, 6,12 and 24 months post surgery
  It is a function of tight muscles weakness that assess the patient inability to achieve the final 15 degrees of active knee extension.
  The therapist/assessor will evaluate if the patient can extend the knee fully with help (passive movement), but have limited range of movement when perform an active knee extension.
  The therapist/assessor will record the degree of limitation for each patient.
  uses a goniometer (instrument that measures an angle of a joint) to measure the degree of knee flexion and extension of a patient.
  Knee Flexion - the measurable degree in which the leg (and knee joint) is bent. Knee Extension - The measurable degree in which the knee is extended (making the joint angle larger, or straightening the knee)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Khoshbin, MD, Principal Investigator — St Michael's Hospital - Unity Health Toronto; Jesse Wolfstadt, MD, Principal Investigator — Mount Sinai Hospital, University of Toronto
Locations (1):
- St Michael's Hospital - Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heiney JP, Barnett MD, Vrabec GA, Schoenfeld AJ, Baji A, Njus GO. Distal femoral fixation: a biomechanical comparison of trigen retrograde intramedullary (i.m.) nail, dynamic condylar screw (DCS), and locking compression plate (LCP) condylar plate. J Trauma. 2009 Feb;66(2):443-9. doi: 10.1097/TA.0b013e31815edeb8. PMID 19204519
- [Background] Papadopoulos EC, Parvizi J, Lai CH, Lewallen DG. Total knee arthroplasty following prior distal femoral fracture. Knee. 2002 Dec;9(4):267-74. doi: 10.1016/s0968-0160(02)00046-7. PMID 12424033
- [Background] Chen F, Li R, Lall A, Schwechter EM. Primary Total Knee Arthroplasty for Distal Femur Fractures: A Systematic Review of Indications, Implants, Techniques, and Results. Am J Orthop (Belle Mead NJ). 2017 May/Jun;46(3):E163-E171. PMID 28666042
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Stevenson M, Segui-Gomez M, Lescohier I, Di Scala C, McDonald-Smith G. An overview of the injury severity score and the new injury severity score. Inj Prev. 2001 Mar;7(1):10-3. doi: 10.1136/ip.7.1.10. PMID 11289527
- [Background] Marsh JL, Slongo TF, Agel J, Broderick JS, Creevey W, DeCoster TA, Prokuski L, Sirkin MS, Ziran B, Henley B, Audige L. Fracture and dislocation classification compendium - 2007: Orthopaedic Trauma Association classification, database and outcomes committee. J Orthop Trauma. 2007 Nov-Dec;21(10 Suppl):S1-133. doi: 10.1097/00005131-200711101-00001. PMID 18277234
- [Background] Kammerlander C, Riedmuller P, Gosch M, Zegg M, Kammerlander-Knauer U, Schmid R, Roth T. Functional outcome and mortality in geriatric distal femoral fractures. Injury. 2012 Jul;43(7):1096-101. doi: 10.1016/j.injury.2012.02.014. Epub 2012 Mar 8. PMID 22405338
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] Wright NC, Looker AC, Saag KG, Curtis JR, Delzell ES, Randall S, Dawson-Hughes B. The recent prevalence of osteoporosis and low bone mass in the United States based on bone mineral density at the femoral neck or lumbar spine. J Bone Miner Res. 2014 Nov;29(11):2520-6. doi: 10.1002/jbmr.2269. PMID 24771492
- [Background] Myers P, Laboe P, Johnson KJ, Fredericks PD, Crichlow RJ, Maar DC, Weber TG. Patient Mortality in Geriatric Distal Femur Fractures. J Orthop Trauma. 2018 Mar;32(3):111-115. doi: 10.1097/BOT.0000000000001078. PMID 29462121
- [Background] Smith JR, Halliday R, Aquilina AL, Morrison RJ, Yip GC, McArthur J, Hull P, Gray A, Kelly MB; Collaborative - Orthopaedic Trauma Society (OTS). Distal femoral fractures: The need to review the standard of care. Injury. 2015;46(6):1084-8. doi: 10.1016/j.injury.2015.02.016. Epub 2015 Feb 26. PMID 25840789
- [Background] Larsen P, Ceccotti AA, Elsoe R. High mortality following distal femur fractures: a cohort study including three hundred and two distal femur fractures. Int Orthop. 2020 Jan;44(1):173-177. doi: 10.1007/s00264-019-04343-9. Epub 2019 May 12. PMID 31081515
- [Background] Boureau F, Benad K, Putman S, Dereudre G, Kern G, Chantelot C. Does primary total knee arthroplasty for acute knee joint fracture maintain autonomy in the elderly? A retrospective study of 21 cases. Orthop Traumatol Surg Res. 2015 Dec;101(8):947-51. doi: 10.1016/j.otsr.2015.09.021. Epub 2015 Nov 14. PMID 26589193
- [Derived] DeFrancesco CJ. CORR Insights(R): How Often Do Complications and Mortality Occur After Operatively Treated Periprosthetic Proximal and Distal Femoral Fractures? A Register-based Study. Clin Orthop Relat Res. 2023 Oct 1;481(10):1950-1953. doi: 10.1097/CORR.0000000000002686. Epub 2023 May 2. No abstract available. PMID 37133402